CLINICAL TRIAL: NCT06270160
Title: Tushirikiane-4-Uthabiti (Supporting Each Other For Resilience)
Brief Title: Livelihoods Intervention With Urban Refugee Youth in Kampala, Uganda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KampalaLivelihoodsStudy
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Financial Stress; Social Functioning; Social Skills
MeSH Terms: conditions — Financial Stress; Social Adjustment; Social Skills

STUDY DESIGN:
Intervention Model Description: The intervention arms will be compared to the control arm of the study using a pre- and post-intervention survey. There will also be a follow-up survey after the study is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: HIVST Alone (Experimental): Participants will be provided with HIVST instructions and education from peer navigators, who will also emphasize the importance of receiving a confirmatory test irrespective of HIV positive result. Peer navigators will demonstrate how to use an HIVST kit, including how to 1) open the kit, 2) collect the oral fluid samples, and 3) read the results. In addition to HIVST education, participants will be offered optional pre-test counselling and SMS contact information to connect with their peer navigator. If participants do not want post-test counselling, the PN will follow up within two weeks. If the participants report testing positive, then they will be immediately scheduled for confirmatory testing and enrolled in the support programs at MARPI for young people living with HIV.
  Interventions: Diagnostic Test: HIVST
- Arm 2: HIVST + mHealth (Experimental): Participants in this arm will be enrolled into the HIVST intervention (as described above) as well as mHealth. The mHealth intervention is a 5-week program that includes a: 1) weekly SMS check-in moderated by the peer navigator; 2) weekly themed informational SMS and accompanying questions to enhance engagement; 3) WhatsApp group multi-media sharing with peer navigators. The peer navigator and coordinator will review group discussions weekly to incentivize engagement; 4) participatory comic books. The investigators are collaborating with the WelTel non-profit agency for a supportive SMS intervention. Weekly 2-way supportive messages will automatically be sent on the same weekday with WelTel software to Arm 2+3 participants, who should respond within 48 hours.
  Interventions: Diagnostic Test: HIVST; Device: mHealth
- Arm 3: HIVST + mHealth + Creating Futures Livelihoods program (Experimental): In addition to HIVST and mHealth access, participants in Arm 3 will also be in enrolled in an 8-week Creating Futures program. This manualized program was developed with youth in South Africa and adapted for the Kenyan context (manual is appended). Topics within the Creating Futures program include: 1) introduction and situating self; 2) sustainable and social resources; 3) peer group meeting; 4) education and learning; 5) getting and keeping jobs; 6) income generating activities; 7) saving and coping with shocks; 8) reflection and looking ahead. This intervention aims to help participants think about, and plan for, their futures to assist them in making a living in the long term. Each workshop is facilitated by pairs of peer navigators and runs from 2-4 hours.
  Interventions: Diagnostic Test: HIVST; Device: mHealth; Behavioral: Creating Futures Livelihoods program

INTERVENTIONS:
Diagnostic Test: HIVST — Peer navigators will demonstrate how to use an HIVST kit, including how to 1) open the kit, 2) collect the oral fluid samples, and 3) read the results. In addition to HIVST education, participants will be offered optional pre-test counselling and SMS contact information to connect with their peer navigator. If participants do not want post-test counselling, the PN will follow up within two weeks. If the participants report testing positive, then they will be immediately scheduled for confirmatory testing and enrolled in the support programs at MARPI for young people living with HIV.
Device: mHealth — The investigators are collaborating with the WelTel non-profit agency for a supportive SMS intervention. The WelTel system will manage the SMS intervention on their structured mobile phone platform (all SMS interactions are logged). Weekly 2-way supportive messages will automatically be sent on the same weekday with WelTel software to Arm 2+3 participants. The peer navigator will ask Arm 2+3 participants to respond to the SMS within 48 hours to confirm their wellbeing and will follow-up with non-responders. The Arm 2+3 peer navigators and Research Coordinator will access the server every 24-48 hours to triage and respond to participants who express a problem or need.
  Arms: Arm 2: HIVST + mHealth; Arm 3: HIVST + mHealth + Creating Futures Livelihoods program
Behavioral: Creating Futures Livelihoods program — Creating Futures is a group intervention that aims to help young people build their livelihoods, and was designed for use with youth (18-24) in urban informal settlements in South Africa.
  Arms: Arm 3: HIVST + mHealth + Creating Futures Livelihoods program

SUMMARY:
Displaced and refugee youth in Uganda are more vulnerable to health risks due to financial insecurity. As such, the investigators aim to explore the utility of an intervention aimed at improving livelihoods, called Creating Futures. Creating Futures is a group intervention that aims to help young people build their livelihoods, and was designed for use with youth (18-24) in urban informal settlements in South Africa.

Since there is a dearth of knowledge regarding efficacious interventions in refugee camps/settlements to engage young people in HIV testing and linkage to care, the investigators will harness various health promotion techniques including mHealth, comics, and the Creating Futures livelihoods intervention to address the urgent needs for: 1) HIV testing interventions with refugee/displaced adolescent and young people in Kampala, and 2) innovative HIV self test (HIVST) delivery strategies to increase linkage to confirmatory testing and HIV care. The investigators will conduct a three-arm cluster randomized controlled trial (cRCT) to evaluate the effectiveness of HIVST delivery methods among AYP living in Kampala. The specific objectives are to: Evaluate the feasibility and effectiveness of: 1) HIVST alone; 2) HIVST in combination with mHealth; and 3) HIVST, mHealth and Creating Futures in combination in increasing routine HIV testing, HIV status knowledge, and linkage to confirmatory testing and HIV care. The investigators aim to examine if adding a livelihoods program to HIV self-testing improves HIV prevention outcomes and other facets of well-being among urban refugee youth in Kampala.

DETAILED DESCRIPTION:
As of March 2021, the prevalence of HIV among Ugandan youth aged 15-24 years was estimated at almost 2%, with young women and adolescent girls having an HIV prevalence over three times that of young men and adolescent boys (2.9% vs. 0.8%). The prevalence of HIV among youth living in Kampala's slums is even higher, at an estimated 13.9-37.2%. This high prevalence may be driven by factors such as food scarcity, limited infrastructure, lack of social support, stigma, and gender norms, which may limit the condom negation and use of HIV testing services among youth. Uganda hosts over 1.5 million refugees, 8% of which reside in Kampala, and many living within slums or informal settlements. While the UNAIDS Gap report identified displaced persons and adolescent girls and young women as populations at high-risk for HIV infection, the HIV prevalence among Uganda's refugees is largely unknown due to the lack of standardized surveillance of refugees.

One approach to improve HIV testing among displaced persons in Uganda is through HIV self-testing (HIVST). HIVST involves a person collecting their own specimen (blood or saliva), conducting the test, and interpreting the results. HIVST has the potential to reduce testing barriers such as stigma and privacy, while enhancing confidentiality and convenience, which are important considerations for adolescents and young people. Innovative HIVST delivery strategies are urgently needed to link persons with positive HIVST results to confirmatory testing and HIV care. As such, identifying strategies to promote linkage to HIV care is essential to realize the public health impact of HIVST. Since there is a dearth of knowledge regarding efficacious interventions in refugee camps/settlements to engage young people in HIV testing and linkage to care, the investigators will harness various health promotion techniques including mHealth, comics, and the Creating Futures livelihoods intervention to address the urgent needs for: 1) HIV testing interventions with refugee/displaced adolescent and young people in Kampala, and 2) innovative HIVST delivery strategies to increase linkage to confirmatory testing and HIV care.

The investigators will evaluate the feasibility and effectiveness of: 1) HIVST alone; 2) HIVST in combination with mHealth; and 3) HIVST, mHealth and Creating Futures in combination in increasing routine HIV testing, HIV status knowledge, and linkage to confirmatory testing and HIV care. The investigators aim to examine if adding a livelihoods program to HIV self-testing improves HIV prevention outcomes and other facets of well-being among urban refugee youth in Kampala.

Mobile health (mHealth) can be used to facilitate HIVST adherence among displaced youth through mobile phone (mHealth) reminders. mHealth approaches are germane to low and middle-income countries (LMIC), where cell phone ownership is rising rapidly, but access to health care is often limited. In Uganda, over 13 million persons have access to mobile phones, and data suggest that HIV prevention messages through mobile phones are beneficial to supplement traditional modalities such as schools for adolescents. Educational comics offer a youth-friendly, low-cost, scalable approach for providing education and health promotion on health topics such as HIV, sexually transmitted infections, vaccines, and dementia. Comics have been used to educate both the general population and healthcare providers to improve care and patient experiences, as they are accessible, do not require high levels of literacy, and can encourage participants to envision and share solutions to sexual violence through facilitating dialogue around emotionally difficult and often stigmatized issues.

Creating Futures is a group intervention that aims to help young people build their livelihoods and was designed for use with youth in urban informal settlements in South Africa. Previous researchers have implemented the Creating Futures intervention in South Africa and found that after the intervention, men's earnings increased, women's experiences of intimate partner violence decreased, men and women scored better on gender attitudes, and depression and suicidal thoughts decreased amongst men.

The investigators will conduct a three-arm cluster randomized controlled trial (cRCT) to evaluate the effectiveness of HIVST delivery methods among youth living in Kampala. The five informal settlements in Kampala will be randomized in a 1:1:1 approach to one of the three study arms. The five informal settlements will be grouped into three sites based on close geographic proximity (1: Kabalagala and Kansanga, 2: Katwe and Nsambya, and 3: Rubaga). The investigators used the following criteria to select informal settlements: 1) settlements that host a large number of refugees or displaced persons; 2) communities with similar measures of socioeconomic status, healthcare access, languages, and living conditions; and 3) evidence of a high prevalence of depressive symptoms among urban refugee youth. Participants will be allocated to a study arm based on their informal settlement of residence. Youth living in slums and informal settlements have shared socio-physical environments. As such, except for individual-level outcome data, the investigators will use a cluster-randomized approach to limit challenges posed by experimental contamination and threats to internal validity. Data collection will be performed at baseline, and 3- and 6-months post-intervention implementation.

The investigators are working with study collaborators from Young African Refugees for Integral Development (YARID), a nongovernmental youth refugee organization in Kampala, who have been involved since the initial research question and focus development stage. The study protocol was developed after a formative qualitative research phase (Phase 1), which included semi-structured interviews with peer navigators and other key informants (e.g., refugee health professionals, migrant workers, teen mothers). Refugee youth aged 18-24 years (12: 6 men, 6 women), living in the same informal settlements who are trained in research methods and ethics will act as peer navigators and enroll other youth in the study after obtaining written informed consent. The investigators employed purposive methods to recruit participants, such as word-of-mouth and venue-based sampling at community events and refugee agencies, beginning with participants who belonged to the Tushirkiane cohort and participated in previous trials on HIVST, COVID-19 prevention, and mental health interventions. The investigators will refresh the cohort with additional purposive recruitment of 16- and 17-year-old participants. The use of SMS and WhatsApp reminders from peer navigators and outreach events allows for the continued engagement and retention of study participants.

Data collection will be conducted by research assistants trained by the Ministry of Health in pre- and post-test counselling. Data will be collected using a structured survey accessed via mobile phones or tablets in all study languages via the SurveyCTO app (Dobility). This app houses a secure platform and automatically encrypts data, which are then uploaded with a Secure Sockets Layer (SSL) certificate to a password-protected server. The use of SurveyCTO allows for multilingual and offline data collection with branching logic and consistency checks. All participants are assigned a unique ID number without any personal identifying information to enhance confidentiality.

The analysis and reporting of this study will be conducted following the CONSORT (Consolidated Standards of Reporting Trials) guidelines. The study analyst will be blinded to group allocation. Participant flow (screening, randomization, allocation, follow-up) will be illustrated using a flow diagram. The investigators will report baseline data for all groups summarized using mean (standard deviation) or median (first and third quartiles) for continuous variables and counts and frequencies (percent) for categorical variables. The investigators will use an intention-to-treat approach with a complete data set whereby participants will be analyzed according to their initial group allocation irrespective of whether they received said intervention.

ELIGIBILITY:
Inclusion Criteria:

* Living in one of the five selected Kampala informal settlements (Kabalagala, Kansanga, Katwe, Nsambya, or Rubaga)
* Identify as a displaced person, refugee, or as having a refugee or displaced parent(s)
* Aged 16-25 years
* Own or have daily access to a mobile phone
* Speak French, English, Kirundi, Kinyarwanda, or Swahili

Exclusion Criteria:

* Not living in one of the five selected informal settlements
* Does not identify as a displaced person, refugee, or as having a refugee or displaced parent(s)
* Aged 15 and under or 26 and older
* Does not have access to a mobile phone or shares a phone
* Does not speak one of French, English, Kirundi, Kinyarwanda, or Swahili

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 432 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants engaged in HIV testing | Every 3 months
  The primary outcome measured in this trial is routine (every 3 months) HIV testing uptake as a measure of HIV prevention. Participants will be asked to self-report when their last HIV test occurred and where it was received (i.e., HIVST, clinic, point-of-care).

SECONDARY OUTCOMES:
Number of participants with knowledge of their HIV status | 3- and 6-month follow-up
  Since HIV status is self-reported, the investigators will use multiple steps to overcome challenges of social desirability bias. First, interviewers will ask participants to report their current HIV status at 3- and 6-month follow-up. Second, the trained interviewer will offer participants a voluntary rapid HIV test (Alere). Knowledge of HIV status will be assessed as correct for participants who agree to take the rapid test and correctly report their HIV status. The investigators will also record if participants were willing to take the interviewer administered rapid test.
Number of participants linked to confirmatory HIV testing | 3- and 6-month follow-up
  Participants will be asked if they used their HIVST kit at 3- and 6-month follow-up. For those who affirm use of HIVST kits with a positive test result, the investigators will ask if and where they received a confirmatory test. Participants can receive confirmatory testing without reporting to the interviewer and can submit coupons at MARPI or to local clinics.
Frequency of linkage to HIV care | 3- and 6-month follow-up
  The investigators will ask participants who seroconvert during the study to report the frequency of HIV care services. In addition, participants can present coupons when accessing MARPI or local clinic services.
Brief HIV Knowledge Questionnaire | 3- and 6-month follow-up
  The investigators will use the18-item dichotomous response (true/false) to assess HIV Knowledge. A score of 0 is recorded for 'false' responses and 1 for 'true responses. A higher total score indicates better knowledge of HIV.
Sexual Risk | 3- and 6-month follow-up
  The investigators will assess sexual risk through self-reported measures of consistent condom use (anal, vaginal sex) with regular, causal, and paid sex partners in the past month, as well as the number of sex partners in the past month, condom use self-efficacy, and selling sex in the past 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Young African Refugees for Integral Development, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The final deidentified data set will be available to users who enter a data-sharing agreement with us. Users will need to (1) secure ethics approval from both their institution and the University of Toronto research ethics board; (2) commit to use the data solely for research purposes, and not to identify any individual participant; (3) commit to securing the data using the appropriate computer technology such as encryption; and (4) commit to destroying or returning the data after analyses are complete.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available 12 months after study completion.
Access Criteria: The final deidentified data set will be available to users who enter a data-sharing agreement with us. Users will need to (1) secure ethics approval from both their institution and the University of Toronto research ethics board; (2) commit to use the data solely for research purposes, and not to identify any individual participant; (3) commit to securing the data using the appropriate computer technology such as encryption; and (4) commit to destroying or returning the data after analyses are complete.

REFERENCES:
- [Background] Culbreth R, Swahn MH, Salazar LF, Ametewee LA, Kasirye R. Risk Factors Associated with HIV, Sexually Transmitted Infections (STI), and HIV/STI Co-infection Among Youth Living in the Slums of Kampala, Uganda. AIDS Behav. 2020 Apr;24(4):1023-1031. doi: 10.1007/s10461-019-02444-5. PMID 30825036
- [Background] Swahn MH, Palmier JB, Kasirye R, Yao H. Correlates of suicide ideation and attempt among youth living in the slums of Kampala. Int J Environ Res Public Health. 2012 Feb;9(2):596-609. doi: 10.3390/ijerph9020596. Epub 2012 Feb 16. PMID 22470312
- [Background] Swahn MH, Culbreth R, Salazar LF, Kasirye R, Seeley J. Prevalence of HIV and Associated Risks of Sex Work among Youth in the Slums of Kampala. AIDS Res Treat. 2016;2016:5360180. doi: 10.1155/2016/5360180. Epub 2016 Apr 28. PMID 27239340
- [Background] Baral S, Logie CH, Grosso A, Wirtz AL, Beyrer C. Modified social ecological model: a tool to guide the assessment of the risks and risk contexts of HIV epidemics. BMC Public Health. 2013 May 17;13:482. doi: 10.1186/1471-2458-13-482. PMID 23679953
- [Background] Sawadogo PM, Sia D, Onadja Y, Beogo I, Sangli G, Sawadogo N, Gnambani A, Bassinga G, Robins S, Tchouaket Nguemeleu E. Barriers and facilitators of access to sexual and reproductive health services among migrant, internally displaced, asylum seeking and refugee women: A scoping review. PLoS One. 2023 Sep 14;18(9):e0291486. doi: 10.1371/journal.pone.0291486. eCollection 2023. PMID 37708137
- [Background] Spiegel PB, Bennedsen AR, Claass J, Bruns L, Patterson N, Yiweza D, Schilperoord M. Prevalence of HIV infection in conflict-affected and displaced people in seven sub-Saharan African countries: a systematic review. Lancet. 2007 Jun 30;369(9580):2187-2195. doi: 10.1016/S0140-6736(07)61015-0. PMID 17604801
- [Background] Warren E, Post N, Hossain M, Blanchet K, Roberts B. Systematic review of the evidence on the effectiveness of sexual and reproductive health interventions in humanitarian crises. BMJ Open. 2015 Dec 18;5(12):e008226. doi: 10.1136/bmjopen-2015-008226. PMID 26685020
- [Background] Jewkes R. Comprehensive response to rape needed in conflict settings. Lancet. 2007 Jun 30;369(9580):2140-2141. doi: 10.1016/S0140-6736(07)60991-X. No abstract available. PMID 17604782
- [Background] Rubenstein BL, Stark L. The impact of humanitarian emergencies on the prevalence of violence against children: an evidence-based ecological framework. Psychol Health Med. 2017 Mar;22(sup1):58-66. doi: 10.1080/13548506.2016.1271949. Epub 2017 Jan 9. PMID 28064522
- [Background] Noble E, Ward L, French S, Falb K. State of the Evidence: A Systematic Review of Approaches to Reduce Gender-Based Violence and Support the Empowerment of Adolescent Girls in Humanitarian Settings. Trauma Violence Abuse. 2019 Jul;20(3):428-434. doi: 10.1177/1524838017699601. Epub 2017 Mar 21. PMID 29334024
- [Background] Logie CH, Okumu M, Mwima S, Hakiza R, Irungi KP, Kyambadde P, Kironde E, Narasimhan M. Social ecological factors associated with experiencing violence among urban refugee and displaced adolescent girls and young women in informal settlements in Kampala, Uganda: a cross-sectional study. Confl Health. 2019 Dec 17;13:60. doi: 10.1186/s13031-019-0242-9. eCollection 2019. PMID 31867053
- [Background] O'Laughlin KN, Rabideau DJ, Kasozi J, Parker RA, Bustamante ND, Faustin ZM, Greenwald KE, Walensky RP, Bassett IV. Predictors of HIV infection: a prospective HIV screening study in a Ugandan refugee settlement. BMC Infect Dis. 2016 Nov 23;16(1):695. doi: 10.1186/s12879-016-2021-1. PMID 27881099
- [Background] O'Laughlin KN, Kasozi J, Rabideau DJ, Parker RA, Mulogo E, Faustin ZM, Greenwald KE, Doraiswamy S, Walensky RP, Bassett IV. The cascade of HIV care among refugees and nationals in Nakivale Refugee Settlement in Uganda. HIV Med. 2017 Aug;18(7):513-518. doi: 10.1111/hiv.12476. Epub 2017 Jan 10. PMID 28070923
- [Background] Pai NP, Thomas R. Time for HIV self-testing in Canada: a vision and an action plan. CMAJ. 2020 Nov 2;192(44):E1367-E1368. doi: 10.1503/cmaj.201160. No abstract available. PMID 33139426
- [Background] Bogart LM, Kgotlaetsile K, Phaladze N, Mosepele M. HIV self-testing may overcome stigma and other barriers to HIV testing among higher-socioeconomic status men in Botswana: A qualitative study. Afr J AIDS Res. 2021 Dec;20(4):297-306. doi: 10.2989/16085906.2021.2000450. PMID 34905451
- [Background] Johnson C, Baggaley R, Forsythe S, van Rooyen H, Ford N, Napierala Mavedzenge S, Corbett E, Natarajan P, Taegtmeyer M. Realizing the potential for HIV self-testing. AIDS Behav. 2014 Jul;18 Suppl 4:S391-5. doi: 10.1007/s10461-014-0832-x. PMID 24986599
- [Background] Hawk ME, Chung A, Creasy SL, Egan JE. A Scoping Review of Patient Preferences for HIV Self-Testing Services in the United States: Implications for Harm Reduction. Patient Prefer Adherence. 2020 Dec 2;14:2365-2375. doi: 10.2147/PPA.S251677. eCollection 2020. PMID 33293799
- [Background] Catania JA, Dolcini MM, Harper GW, Dowhower DP, Dolcini-Catania LG, Towner SL, Timmons A, Motley DN, Tyler DH. Bridging barriers to clinic-based HIV testing with new technology: translating self-implemented testing for African American youth. Transl Behav Med. 2015 Dec;5(4):372-83. doi: 10.1007/s13142-015-0331-2. Epub 2015 Jun 9. PMID 26622910
- [Background] Brown W 3rd, Carballo-Dieguez A, John RM, Schnall R. Information, Motivation, and Behavioral Skills of High-Risk Young Adults to Use the HIV Self-Test. AIDS Behav. 2016 Sep;20(9):2000-9. doi: 10.1007/s10461-016-1309-x. PMID 26885813
- [Background] Choko AT, MacPherson P, Webb EL, Willey BA, Feasy H, Sambakunsi R, Mdolo A, Makombe SD, Desmond N, Hayes R, Maheswaran H, Corbett EL. Uptake, Accuracy, Safety, and Linkage into Care over Two Years of Promoting Annual Self-Testing for HIV in Blantyre, Malawi: A Community-Based Prospective Study. PLoS Med. 2015 Sep 8;12(9):e1001873. doi: 10.1371/journal.pmed.1001873. eCollection 2015 Sep. PMID 26348035
- [Background] Johnson CC, Kennedy C, Fonner V, Siegfried N, Figueroa C, Dalal S, Sands A, Baggaley R. Examining the effects of HIV self-testing compared to standard HIV testing services: a systematic review and meta-analysis. J Int AIDS Soc. 2017 May 15;20(1):21594. doi: 10.7448/IAS.20.1.21594. PMID 28530049
- [Background] Cambiano V, Mavedzenge SN, Phillips A. Modelling the potential population impact and cost-effectiveness of self-testing for HIV: evaluation of data requirements. AIDS Behav. 2014 Jul;18 Suppl 4(Suppl 4):S450-8. doi: 10.1007/s10461-014-0824-x. PMID 24957978
- [Background] Govindasamy D, Meghij J, Kebede Negussi E, Clare Baggaley R, Ford N, Kranzer K. Interventions to improve or facilitate linkage to or retention in pre-ART (HIV) care and initiation of ART in low- and middle-income settings--a systematic review. J Int AIDS Soc. 2014 Aug 1;17(1):19032. doi: 10.7448/IAS.17.1.19032. eCollection 2014. PMID 25095831
- [Background] Logie CH, Okumu M, Berry I, Hakiza R, Baral SD, Musoke DK, Nakitende A, Mwima S, Kyambadde P, Loutet M, Batte S, Lester R, Neema S, Newby K, Mbuagbaw L. Findings from the Tushirikiane mobile health (mHealth) HIV self-testing pragmatic trial with refugee adolescents and youth living in informal settlements in Kampala, Uganda. J Int AIDS Soc. 2023 Oct;26(10):e26185. doi: 10.1002/jia2.26185. PMID 37850816
- [Background] Mitchell KJ, Bull S, Kiwanuka J, Ybarra ML. Cell phone usage among adolescents in Uganda: acceptability for relaying health information. Health Educ Res. 2011 Oct;26(5):770-81. doi: 10.1093/her/cyr022. Epub 2011 May 2. PMID 21536715
- [Background] Twimukye A, Bwanika Naggirinya A, Parkes-Ratanshi R, Kasirye R, Kiragga A, Castelnuovo B, Wasswa J, Nabaggala MS, Katabira E, Lamorde M, King RL. Acceptability of a Mobile Phone Support Tool (Call for Life Uganda) for Promoting Adherence to Antiretroviral Therapy Among Young Adults in a Randomized Controlled Trial: Exploratory Qualitative Study. JMIR Mhealth Uhealth. 2021 Jun 14;9(6):e17418. doi: 10.2196/17418. PMID 34121665
- [Background] Shin MB, Ko LK, Ibrahim A, Mohamed FB, Lin J, Celentano I, Shankar M, Amsalu F, Ali AA, Richardson BA, Taylor VM, Winer RL. The Impact of a Comic Book Intervention on East African-American Adolescents' HPV Vaccine-Related Knowledge, Beliefs and Intentions. J Immigr Minor Health. 2022 Dec;24(6):1489-1500. doi: 10.1007/s10903-022-01359-z. Epub 2022 Mar 31. PMID 35357620
- [Background] Tekle-Haimanot R, Preux PM, Gerard D, Worku DK, Belay HD, Gebrewold MA. Impact of an educational comic book on epilepsy-related knowledge, awareness, and attitudes among school children in Ethiopia. Epilepsy Behav. 2016 Aug;61:218-223. doi: 10.1016/j.yebeh.2016.05.002. Epub 2016 Jul 1. PMID 27372962
- [Background] Vujcich D, Thomas J, Crawford K, Ward J. Indigenous Youth Peer-Led Health Promotion in Canada, New Zealand, Australia, and the United States: A Systematic Review of the Approaches, Study Designs, and Effectiveness. Front Public Health. 2018 Feb 13;6:31. doi: 10.3389/fpubh.2018.00031. eCollection 2018. PMID 29497608
- [Background] Muzumdar JM, Pantaleo NL. Comics as a Medium for Providing Information on Adult Immunizations. J Health Commun. 2017 Oct;22(10):783-791. doi: 10.1080/10810730.2017.1355418. Epub 2017 Sep 13. PMID 28901823
- [Background] Krasnoryadtseva A, Dalbeth N, Petrie KJ. The effect of different styles of medical illustration on information comprehension, the perception of educational material and illness beliefs. Patient Educ Couns. 2020 Mar;103(3):556-562. doi: 10.1016/j.pec.2019.09.026. Epub 2019 Sep 27. PMID 31601448
- [Background] Gallagher-Thompson D, Tzuang M, Hinton L, Alvarez P, Rengifo J, Valverde I, Chen N, Emrani T, Thompson LW. Effectiveness of a fotonovela for reducing depression and stress in Latino dementia family caregivers. Alzheimer Dis Assoc Disord. 2015 Apr-Jun;29(2):146-53. doi: 10.1097/WAD.0000000000000077. PMID 25590939
- [Background] Towey F. Conference: Comics and medicine. Lancet Oncol. 2014 Aug;15(9):927-8. doi: 10.1016/s1470-2045(14)70352-3. No abstract available. PMID 25225688
- [Background] Waite M. Writing medical comics. J Vis Commun Med. 2019 Jul;42(3):144-150. doi: 10.1080/17453054.2019.1575641. Epub 2019 Aug 8. PMID 31394951
- [Background] Unger JB, Cabassa LJ, Molina GB, Contreras S, Baron M. Evaluation of a fotonovela to increase depression knowledge and reduce stigma among Hispanic adults. J Immigr Minor Health. 2013 Apr;15(2):398-406. doi: 10.1007/s10903-012-9623-5. PMID 22485012
- [Background] Misselhorn A, Mushinga M, Jama-Shai N, Washington L, Mbatha M. Creating Futures: Supporting Young People in Building their Livelihoods. Health Economics and HIV and AIDS Research Division (HEARD), University of KwaZulu-Natal. 2013.
- [Background] Jewkes R, Gibbs A, Jama-Shai N, Willan S, Misselhorn A, Mushinga M, Washington L, Mbatha N, Skiweyiya Y. Stepping Stones and Creating Futures intervention: shortened interrupted time series evaluation of a behavioural and structural health promotion and violence prevention intervention for young people in informal settlements in Durban, South Africa. BMC Public Health. 2014 Dec 29;14:1325. doi: 10.1186/1471-2458-14-1325. PMID 25544716
- [Background] Embleton L, Di Ruggiero E, Logie CH, Ayuku D, Braitstein P. Improving livelihoods and gender equitable attitudes of street-connected young people in Eldoret, Kenya: Results from a pilot evidence-based intervention. Health Soc Care Community. 2021 Jan;29(1):227-240. doi: 10.1111/hsc.13086. Epub 2020 Jul 7. PMID 32633059
- [Background] Embleton L, Di Ruggiero E, Odep Okal E, Chan AK, Logie CH, Ayuku D, Braitstein P. Adapting an evidence-based gender, livelihoods, and HIV prevention intervention with street-connected young people in Eldoret, Kenya. Glob Public Health. 2019 Dec;14(12):1703-1717. doi: 10.1080/17441692.2019.1625940. Epub 2019 Jun 4. PMID 31162989
- [Background] Logie CH, Okumu M, Kortenaar JL, Gittings L, Khan N, Hakiza R, Kibuuka Musoke D, Nakitende A, Katisi B, Kyambadde P, Khan T, Lester R, Mbuagbaw L. Mobile Health-Supported Virtual Reality and Group Problem Management Plus: Protocol for a Cluster Randomized Trial Among Urban Refugee and Displaced Youth in Kampala, Uganda (Tushirikiane4MH, Supporting Each Other for Mental Health). JMIR Res Protoc. 2022 Dec 8;11(12):e42342. doi: 10.2196/42342. PMID 36480274
- [Background] Lyytinen E. Informal places of protection: Congolese refugees' 'communities of trust' in Kampala, Uganda. Journal of Ethnic and Migration Studies. 2017 Apr 26;43(6):991-1008.
- [Background] Logie CH, Berry I, Okumu M, Loutet M, McNamee C, Hakiza R, Musoke DK, Mwima S, Kyambadde P, Mbuagbaw L. The prevalence and correlates of depression before and after the COVID-19 pandemic declaration among urban refugee adolescents and youth in informal settlements in Kampala, Uganda: A longitudinal cohort study. Ann Epidemiol. 2022 Feb;66:37-43. doi: 10.1016/j.annepidem.2021.11.005. Epub 2021 Nov 14. PMID 34785396
- [Background] Logie CH, Okumu M, Mwima S, Hakiza R, Chemutai D, Kyambadde P. Contextual factors associated with depression among urban refugee and displaced youth in Kampala, Uganda: findings from a cross-sectional study. Confl Health. 2020 Jul 10;14:45. doi: 10.1186/s13031-020-00289-7. eCollection 2020. PMID 32665785
- [Background] Logie C, Okumu M, Hakiza R, Kibuuka Musoke D, Berry I, Mwima S, Kyambadde P, Kiera UM, Loutet M, Neema S, Newby K, McNamee C, Baral SD, Lester R, Musinguzi J, Mbuagbaw L. Mobile Health-Supported HIV Self-Testing Strategy Among Urban Refugee and Displaced Youth in Kampala, Uganda: Protocol for a Cluster Randomized Trial (Tushirikiane, Supporting Each Other). JMIR Res Protoc. 2021 Feb 2;10(2):e26192. doi: 10.2196/26192. PMID 33528378
- [Background] Logie CH, Okumu M, Berry I, Hakiza R, Kibuuka Musoke D, Kyambadde P, Mwima S, Lester RT, Perez-Brumer AG, Baral S, Mbuagbaw L. Kukaa Salama (Staying Safe): study protocol for a pre/post-trial of an interactive mHealth intervention for increasing COVID-19 prevention practices with urban refugee youth in Kampala, Uganda. BMJ Open. 2021 Nov 22;11(11):e055530. doi: 10.1136/bmjopen-2021-055530. PMID 34810193
- [Background] Carey MP, Schroder KE. Development and psychometric evaluation of the brief HIV Knowledge Questionnaire. AIDS Educ Prev. 2002 Apr;14(2):172-82. doi: 10.1521/aeap.14.2.172.23902. PMID 12000234
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Bland JM, Altman DG. Multiple significance tests: the Bonferroni method. BMJ. 1995 Jan 21;310(6973):170. doi: 10.1136/bmj.310.6973.170. No abstract available. PMID 7833759
- [Background] Schober P, Vetter TR. Adjustments for Multiple Testing in Medical Research. Anesth Analg. 2020 Jan;130(1):99. doi: 10.1213/ANE.0000000000004545. No abstract available. PMID 31842175
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Derived] Logie CH, Okumu M, Tailor L, MacKenzie F, Admassu Z, Hakiza R, Kibuuka Musoke D, Katisi B, Nakitende A, Kyambadde P, Mbuagbaw L. Tushirikiane-4-Uthabiti (Supporting Each Other For Resilience): study protocol of a mental health, HIV self-testing and livelihoods randomised controlled trial for advancing HIV prevention outcomes among urban refugee youth in Kampala, Uganda. BMJ Open. 2024 Nov 24;14(11):e087470. doi: 10.1136/bmjopen-2024-087470. PMID 39581739
- See also: Uganda Population-Based HIV Impact Assessment 2020 — https://phia.icap.columbia.edu/wp-content/uploads/2022/08/UPHIA-Summary-Sheet-2020.pdf
- See also: UNAIDS 90-90-90: An Ambitious Treatment Target to Help End the AIDS Epidemic — http://www.unaids.org/sites/default/files/media_asset/90-90-90_en.pdf
- See also: UN General Assembly resoluation: Political Declaration on HIV and AIDS: On the Fast-Track to Accelerate the Fight against HIV and to End the AIDS Epidemic by 2030 — http://www.unaids.org/sites/default/files/media_asset/2016-political-declaration-HIV-AIDS_en.pdf
- See also: UNAIDS: A Super-Fast-Track Framework for Ending AIDS among Children, Adolescent and Young Women by 2020 — http://www.unaids.org/sites/default/files/media_asset/Stay_free_vision_mission_En.pdf
- See also: Refugee Statistics — https://www.unrefugees.org/refugee-facts/statistics/
- See also: Overview of Refugees and Asylum-seekers in Uganda — https://reporting.unhcr.org/operational/operations/uganda#:~:text=Most%20refugees%20come%20from%20South,additional%208%25%20reside%20in%20Kampala.
- See also: Urban Refugees: Kampala, Uganda — http://www.urban-refugees.org/kampala/
- See also: Refugee livelihoods in Kampala, Nakivale and Kyangwali refugee settlements Patterns of engagement with the private sector. — http://www.rsc.ox.ac.uk/files/publications/working-paper-series/wp95-refugee-livelihoods-kampala-nakivale-kyangwali-2013.pdf
- See also: UNAIDS: HIV Gap Report — https://www.unaids.org/en/resources/campaigns/2014/2014gapreport/gapreport
- See also: Insights into potential users and messaging for HIV oral self-test kits in Kenya — https://www.3ieimpact.org/sites/default/files/2018-12/insights_into_potential_users-final.pdf
- See also: mHealth: New horizons for health through mobile technologies — http://www.webcitation.org/63mBxLED9
- See also: COVID-19 socioeconomic impact worsens for refugees in Uganda — https://www.unhcr.org/blogs/https-www-unhcr-org-blogs-covid-19-socioeconomic-impact-worsens-for-refugees-in-uganda/